CLINICAL TRIAL: NCT00756223
Title: An Open-label Phase I Single Dose Escalation Trial of Two Dosing Schedules of BI 831266 Administered Intravenously Over 24 h Continuously in Patients With Advanced Solid Tumours
Brief Title: Phase I Study of BI 831266 in Patients With Advanced Solid Tumours
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1257.1; 2008-001631-36 (EudraCT Number: EudraCT)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Last update posted 2013-11-21 (Estimated); Status verified 2013-11

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

ARMS (2):
- Arm A (Experimental): BI 831266 24h infusion on day 1 and day 15 every 4 weeks
  Interventions: Drug: Arm A
- Arm B (Experimental): BI 831266 24h infusion on day 1 every 3 weeks
  Interventions: Drug: Arm B

INTERVENTIONS:
Drug: Arm A — Dose escalation Arm A (4 weeks)
  Arms: Arm A
Drug: Arm B — Dose escalation Arm B (3 weeks)
  Arms: Arm B

SUMMARY:
The main objective of this trial is to provide safety data in terms of drug-related adverse events for the recommendation of the dose for further trials in the development of BI 831266.

Secondary objectives are the collection of antitumour efficacy data and the determination of the pharmacokinetic and pharmacodynamic profile of BI 831266.

ELIGIBILITY:
Inclusion criteria:

1. Patients with confirmed diagnosis of advanced, non-resectable and/or metastatic solid malignant tumours, who have failed conventional treatment or for whom no therapy of proven efficacy exists or who are not amenable to established treatment options
2. Secure central venous access
3. Measurable and/or non-measurable tumour deposits
4. Recovery from toxicities of prior anti-cancer therapies at least to CTCAE grade 1
5. Age >= 18 years
6. Life expectancy >= 3 months
7. Written informed consent in accordance with International Conference on Harmonisation guideline for Good Clinical Practice and local legislation
8. Eastern Cooperative Oncology Group performance score <= 2

Exclusion criteria:

1. Serious illness, concomitant non-oncological disease (e.g. active infectious disease), or ongoing toxicity of prior therapies considered by the investigator to potentially compromise patients' safety in this trial
2. Pregnancy or breastfeeding
3. Symptomatic brain metastases and/or leptomeningeal disease requiring therapy
4. Second malignancy requiring therapy
5. Left ventricular ejection fraction (LVEF) < 50% in echocardiography
6. Clinically significant (i.e. active) cardiovascular disease: CVA/stroke (<= 6 months prior to randomisation), myocardial infarction (<= 6 months prior to randomisation), unstable angina, New York Heart Association Grade II or greater congestive heart failure, or serious cardiac arrhythmia requiring medication
7. Absolute neutrophil count less than 1500 / mm3
8. Platelet count less than 100 000 / mm3
9. Bilirubin greater than 1.5 mg / dl (> 26 micromol / L, SI unit equivalent)
10. Aspartate amino transferase (AST) and / or alanine amino transferase (ALT) greater than 2.5 times the upper limit of normal (if related to liver metastases greater than five times the upper limit of normal)
11. Serum creatinine greater than 1.5 mg / dl (> 132 micromol / L, SI unit equivalent)
12. Women and men who are sexually active and unwilling to use a medically acceptable method of contraception
13. Treatment with other investigational drugs or in another clinical trial within the past two weeks before start of therapy or concomitantly with this trial
14. Chemo-, hormone, radio- or immunotherapy within the past two weeks before start of therapy or concomitantly with this trial
15. Patients unable to comply with the protocol
16. Active alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2008-11; Primary Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose | 3-4 weeks

SECONDARY OUTCOMES:
Safety parameters (incidence and intensity of AEs graded according to the common terminology criteria for AEs and incidence of DLT) | throughout the study period
Pharmacokinetic parameters | throughout the study period
Pharmacodynamic analysis | 3-4 weeks
Efficacy data (progression free survival, objective response rate, response duration) | throughout the study period

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (3):
- Austria (3):
  - 1257.1.4303 Boehringer Ingelheim Investigational Site, Linz
  - 1257.1.4302 Boehringer Ingelheim Investigational Site, Salzburg
  - 1257.1.4301 Boehringer Ingelheim Investigational Site, Vienna

REFERENCES:
- [Derived] Dittrich C, Fridrik MA, Koenigsberg R, Lee C, Goeldner RG, Hilbert J, Greil R. A phase 1 dose escalation study of BI 831266, an inhibitor of Aurora kinase B, in patients with advanced solid tumors. Invest New Drugs. 2015 Apr;33(2):409-22. doi: 10.1007/s10637-014-0201-7. Epub 2014 Dec 23. PMID 25529193